CLINICAL TRIAL: NCT01986972
Title: Supragingival Plaque Removal With and Without Dentifrice: A Randomized Controlled Trial
Brief Title: Supragingival Plaque Removal With and Without Dentifrice
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Franciscan University Center (Other)
Responsible Party: Principal Investigator, Raquel Pippi Antoniazzi, Supragingival Plaque Removal With and Without Dentifrice: A Randomized Controlled Trial, Franciscan University Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: RAntoniazzi
Record Dates: First submitted 2013-03-09; First posted 2013-11-19 (Estimated); Last update posted 2013-11-19 (Estimated); Status verified 2013-11

CONDITIONS: Dental Plaque
Keywords: Toothbrushing; Dental plaque; Dentifrice; Oral hygiene
MeSH Terms: conditions — Dental Plaque | interventions — Toothbrushing; Dentifrices

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Toothbrushing With Dentifrice (Active Comparator): After 72 hours of absence oral hygiene, patients performed toothbrushing with common dentifrice.
  Interventions: Other: Toothbrushing With Dentifrice
- Toothbrushing Without Dentifrice (Experimental): After 72 hours of absence oral hygiene, patients performed toothbrushing without dentifrice.
  Interventions: Other: Toothbrushing Without Dentifrice

INTERVENTIONS:
Other: Toothbrushing With Dentifrice — The participants were instructed to interrupt any chemical and/or mechanical oral hygiene procedure for 72 hours. Dental plaque was stained by a 2% erithrosin solution, followed by a mouth rinsing with water for 1 minute. Next, the set of dental quadrants (1-3 and 2-4) were randomly allocated to experimental groups by the flip of a coin. One of the sets was brushed with multi bristle brush without the use of dentifrice and the second set was brushed with multi bristle brush using dentifrice. Toothbrushing was performed by the individual's regular technique timed. Two minutes was used for each set. After toothbrushing, the dental biofilm was again stained and evaluated by the same examiner, who was blind to the quadrants brushed with or without dentifrice.
  Other Names: Brushed with multi bristle brush; Dentifrice closeUp
  Arms: Toothbrushing With Dentifrice
Other: Toothbrushing Without Dentifrice — The participants were instructed to interrupt any chemical and/or mechanical oral hygiene procedure for 72 hours. Then, dental plaque was stained by a 2% erithrosin solution, followed by a mouth rinsing with water for 1 minute. Next, the set of dental quadrants (1-3 and 2-4) were randomly allocated to experimental groups by the flip of a coin. One of the sets was brushed with multi bristle brush without the use of dentifrice and the second set was brushed with multi bristle brush using dentifrice. Toothbrushing was performed by the individual's regular technique timed. Two minutes was used for each set. After toothbrushing, the dental biofilm was again stained and evaluated by the same examiner, who was blind to the quadrants brushed with or without dentifrice.
  Arms: Toothbrushing Without Dentifrice

SUMMARY:
Purpose: The aim of this study was to compare the efficacy of dental biofilm removal by brushing with and without conventional toothpaste. Settings and Design: Twenty-four students aged 17 to 28 years old participated in this randomized clinical trial.

Materials and Methods: Quadrants 1-3 or 2-4 were randomly allocated to the test group (brushing without dentifrice) or control group (brushing with dentifrice). After 72 hours of cessation of oral hygiene, Quigley & Hein (Turesky) plaque index was assessed before and after brushing by a calibrated and blind examiner. Overtime and intergroup comparisons were performed by paired sample t test.

ELIGIBILITY:
Inclusion Criteria:

* students of both genders systemically healthy.

Exclusion Criteria:

* individuals who exhibited gingivitis (presence of gingival bleeding at any site);
* probing depth > 3mm and/or attachment loss >3mm at any site;
* using orthodontic appliance devices, dental prostheses, dental implants;
* presence of abrasions, restorations and/or carious lesions at cervical region;
* individuals who had less than 20 natural teeth.

Ages: 17 Years to 28 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2009-07; Primary Completion 2010-09 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Dental plaque | Three days
  The presence of plaque was determined by Quigley and Hein (QH) (19) modified by Turesky index.

CONTACTS AND LOCATIONS:
Locations (1):
- School of Dentistry, Franciscan University Center, Santa Maria, Rio Grande do Sul, Brazil